CLINICAL TRIAL: NCT05665387
Title: OPSIS: A Phase IIa, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, Multicenter Study Assessing the Efficacy and Safety of STN1013600 Ophthalmic Solution 0.1% and 0.3% Compared With Placebo in Subjects With Presbyopia
Brief Title: Study Assessing the Efficacy and Safety of STN1013600 Ophthalmic Solution 0.1% and 0.3% Compared With Placebo in Subjects With Presbyopia
Acronym: OPSIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101360002IN
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Presbyopia
Keywords: Santen, Presbyopia, Eye
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.1% STN1013600 ophthalmic solution (Experimental): 0.1% STN1013600 ophthalmic solution 1 drop BID
  Interventions: Drug: 0.1% STN1013600 ophthalmic solution
- 0.3% STN1013600 ophthalmic solution (Experimental): 0.3% STN1013600 ophthalmic solution 1 drop BID
  Interventions: Drug: 0.3% STN1013600 ophthalmic solution
- Placebo (Vehicle) ophthalmic solution (Placebo Comparator): Placebo (Vehicle) ophthalmic solution BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.1% STN1013600 ophthalmic solution — 0.1% STN1013600 ophthalmic solution 1 drop BID for 2 months
  Arms: 0.1% STN1013600 ophthalmic solution
Drug: 0.3% STN1013600 ophthalmic solution — 0.3% STN1013600 ophthalmic solution 1 drop BID for 2 months
  Arms: 0.3% STN1013600 ophthalmic solution
Drug: Placebo — Placebo ophthalmic solution 1 drop BID for 2 months
  Arms: Placebo (Vehicle) ophthalmic solution

SUMMARY:
This is a Phase IIa study to assess efficacy and safety of STN1013600 ophthalmic solution (0.1%, and 0.3 %), twice daily when compared to Placebo in subjects diagnosed with presbyopia. This study will consist of a Screening Period of up to 15 days followed by a 2 Month Treatment Period. After the Treatment Period subjects will be followed for a one-month treatment free period.

ELIGIBILITY:
Inclusion Criteria:

* Phakic presbyopic subjects, Male or Female between 47 and 55 years of age.
* Distance-corrected near visual acuity (DCNVA) for each eye, as well as for binocular vision, 70 EDTRS letters or worse (equivalent to 0.3 logMAR or worse; or 20/40 Snellen or worse) at 40 cm. To be reconfirmed at Visit 2 (Baseline).
* Best-corrected distance visual acuity (BCDVA) for each eye of 85 ETDRS letters or better (equivalent to 0.00 logMAR or better; or 20/20 Snellen or better) at 4 m. To be reconfirmed at Visit 2 (Baseline).

Exclusion Criteria:

* Secondary cause of presbyopia in either eye as assessed by investigator (e.g., damage to lens, zonules or ciliary muscle, multiple sclerosis, cardiovascular accidents, vascular insufficiency, myasthenia gravis, anemia, influenza, measles).
* Any history of ocular surgery (including ocular laser surgery) in either eye or plan of ocular surgery (including ocular laser surgery) during the course of the study.
* Prior invasive therapy for presbyopia (e.g., ciliary body electrostimulation, corneal implants).

Ages: 47 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Global Research Management Inc, Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Comprehensive Eye Care, Ltd, Washington, Missouri
  - Rochester Ophthalmological Group, P.C., Rochester, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - Scott Christie and Associates PC, Cranberry Township, Pennsylvania
  - Vance Thompson Vision Clinic, Sioux Falls, South Dakota
  - University Eye Specialists, Maryville, Tennessee
  - Total Eye Care PA, Memphis, Tennessee
  - The Cataract and Glaucoma Center, El Paso, Texas
  - R and R Eye Research LLC, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Started | 30 | 33 | 16
Completed | 29 | 33 | 15
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution | Total
Number analyzed (Participants) | 30 | 33 | 16 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 16 | 79
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (2.20) | 51.1 (2.51) | 51.4 (1.78) | 51.4 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 11 | 50
  Male | 13 | 11 | 5 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 0 | 11
  White | 27 | 23 | 14 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 16 | 79

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Binocular Distance Corrected Near Visual Acuity (DCNVA)
Description: Analysis of Change from Baseline at Month 2 was done using Bayesian Approach Analysis Population.
Time Frame: At Month 2
Population: Full Analysis Set (FAS) included all randomized subjects. The number analyzed are participants evaluable for the outcome measure at Month 2.
Measure: Mean (Standard Error); unit: EDTRS letters
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Number analyzed (Participants) | 30 | 33 | 15
EDTRS letters | 4.1 (1.24) | 4.3 (1.18) | 4.4 (1.13)

2. Secondary Outcome: Mean Change From Baseline in Study Eye Distance Corrected Near Visual Acuity (DCNVA) at Month 2
Description: Summary of Early Treatment Diabetic Retinopathy Study (ETDRS) Letters and Change from Baseline by Analysis Visit.
Time Frame: Month 2
Population: Full Analysis Set (observed cases only).
Measure: Mean (Standard Deviation); unit: EDTRS letters
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Number analyzed (Participants) | 30 | 33 | 15
EDTRS letters
  Baseline Observed | 62.2 (6.29) | 63.5 (4.84) | 63.8 (4.71)
  Month 2 Observed | 66.4 (6.69) | 67.9 (8.10) | 68.7 (7.58)
  Month 2 Change from Baseline | 4.2 (6.65) | 4.4 (7.15) | 4.8 (5.88)

3. Secondary Outcome: Percentage of Participants Who Improved 1/2/3-lines or More in Study Eye and Binocular Distance Corrected Near Visual Acuity (DCNVA) at Month 2
Description: The response rate is the percentage of participants that achieved the specified gain in Distance Corrected Intermediate Visual Acuity (DCIVA) without losing more than 5 ETDRS (Early Treatment Diabetic Retinopathy Study) letters in Best Corrected Distance Visual Acuity (BCDVA)
Time Frame: Month 2
Population: Full Analysis Set (observed cases only).
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Number analyzed (Participants) | 30 | 33 | 15
Participants
  Month 2 Having a gain of 5 or more letters in DCIVA without loosing more than 5 letters in BCDVA | 13 | 17 | 5
  Month 2 Having a gain of 10 or more letters in DCIVA without loosing more than 5 letters in BCDVA | 6 | 12 | 0
  Month 2 Having a gain of 15 or more letters in DCIVA without loosing more than 5 letters in BCDVA | 1 | 5 | 0

4. Secondary Outcome: Mean Change From Baseline in Quality of Life Assessed With Near Activity Visual Questionnaire (NAVQ) at Month 2
Description: Analysis of change from baseline in Rasch Score was done using Mixed-Effects Model for Repeated Measures (MMRM). Least Square Means were obtained by fitting a MMRM model to the NAVQ values.
  The summated NAVQ score from initial 10 questions ranged from 0 to 30, where higher score indicates more difficulty with near tasks. The summated NAVQ score is converted to Rasch score which ranged from 0 to 100, with higher values indicating more difficulty with near tasks.
Time Frame: Month 2
Population: Full Analysis Set (observed cases only).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Number analyzed (Participants) | 30 | 33 | 15
score on a scale | -7.493 (2.1803) | -8.140 (2.0939) | -10.510 (3.1447)

5. Secondary Outcome: Subject Treatment Satisfaction as Assessed by Patient Global Rating of Treatment
Description: The response rate is the percent of participants that responded with "Satisfactory" or "Very Satisfactory" when asked to rate the overall satisfaction with the treatment.
Time Frame: Month 2
Population: Full Analysis Set (Observed cases only)
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
Number analyzed (Participants) | 30 | 33 | 15
Participants | 13 | 18 | 9

ADVERSE EVENTS:
Time Frame: Adverse events in this study were collected from the time of informed consent and until subject withdrawal or until the subject's participation in the study ended at 3 Months.
Description: Reported AEs were followed by the investigator until resolution, stabilization, the event was otherwise explained, or the participant is lost to follow up.
Arm/Group | 0.3% STN1013600 Ophthalmic Solution | 0.1% STN1013600 Ophthalmic Solution | Placebo (Vehicle) Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33 | 0/16
Other Adverse Events (participants affected / at risk) | 7/30 | 9/33 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% STN1013600 Ophthalmic Solution (N=30) | 0.1% STN1013600 Ophthalmic Solution (N=33) | Placebo (Vehicle) Ophthalmic Solution (N=16)
Eye irritation (Eye disorders) | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Instillation site irritation (General disorders) | 1 | 2 | 0
Instillation site discomfort (General disorders) | 1 | 0 | 0
Liver function test increased (Investigations) | 1 | 2 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT05665387/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05665387/SAP_001.pdf